CLINICAL TRIAL: NCT01469520
Title: Phase I Three-way Crossover Bioequivalence Study of Pediatric Formulations of Lamivudine/Zidovudine/Nevirapine Using Healthy Adult Volunteers
Brief Title: Bioequivalence Study of Pediatric Formulations to Treat HIV Infection
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Elim Pediatric Pharmaceuticals Inc. (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: RU 2010-73; 2010-73 (Other: Roosevelt University)
Record Dates: First submitted 2011-11-04; First posted 2011-11-10 (Estimated); Last update posted 2011-11-10 (Estimated); Status verified 2011-11

CONDITIONS: HIV; AIDS
Keywords: HIV; AIDS; Treatment
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome | interventions — Lamivudine; Zidovudine; Nevirapine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Reference (Active Comparator): Co-administered liquid mixture of Epivir® (lamivudine) solution, Retrovir® (zidovudine)and Viramune® (nevirapine)
  Interventions: Drug: Epivir®, Retrovir® and Viramune®
- Test product (Active Comparator): Fixed dose combination of lamivudine, zidovudine and nevirapine reconstitutable suspension
  Interventions: Drug: Lamivudine, Zidovudine and nevirapine; Drug: Lamivudine, zidovudine, nevirapine
- Test Product (Active Comparator): Fixed dose combination combination (Lamivudine, Zidovudine and Nevirapine)tablet
  Interventions: Drug: Lamivudine, Zidovudine and nevirapine; Drug: Lamivudine, zidovudine, nevirapine

INTERVENTIONS:
Drug: Epivir®, Retrovir® and Viramune® — 12 mL of Epivir® (lamivudine) 10 mg/mL solution plus 24 ml of Retrovir® (zidovudine) 10 mg/mL syrup plus and 20 mL of Viramune® (nevirapine) of 10 mg/mL
  Other Names: Lamivudine; Zidovudine; Nevirapine
  Arms: Reference
Drug: Lamivudine, Zidovudine and nevirapine — 20 mL of reconstituted granules for suspension containing lamivudine 30mg/zidovudine 60 mg/nevirapine 50 mg per 5 mL of suspension
  Other Names: Lamivudine; Zidovudine; Nevirapine
  Arms: Test Product; Test product
Drug: Lamivudine, zidovudine, nevirapine — Lamivudine 30mg/zidovudine 60 mg/nevirapine 50 mg per tablet.
  Other Names: Lamivudine; Zidovudine; Nevirapine
  Arms: Test Product; Test product

SUMMARY:
The purpose of the study is to determine the bioavailability/bioequivalence of two pediatric formulations (tablet and reconstitutable suspension) of lamivudine/zidovudine/ nevirapine in comparison to an innovator product. Establishing the bioequivalence of a newly developed age-appropriate fixed dose combination of lamivudine/zidovudine/ nevirapine as an oral dispersible tablet or a reconstitutable suspension for children is invaluable for future product registration and availability of the products to children, thus filling the void in pediatric HIV/AIDS therapy.

DETAILED DESCRIPTION:
Volunteer Selection and Size: The International Conference on Harmonization (ICH) guideline E11 on clinical investigation of medicinal products in the pediatric population suggests that for relative bioavailability comparison of pediatric formulations, adult subjects may be used. Therefore, the study will be performed in a minimum of 24 healthy adult subjects. However, 29 healthy adults will be enrolled to allow for two possible drop-outs and for three subjects that may develop hypersensitivity to nevirapine which is known for its hypersensitivity side effect, in form of rashes.

In anticipation of such reactions,10% more of the 26 subjects will be added to the group. This will make a total of 29 volunteers during the study. Advertisements announcing the study will be posted at the Bowen University Teaching Hospital two months before the commencement of the study to invite volunteers.

Informed Consent Procedure: The volunteers will be screened using a questionnaire (see attached). The language of communication will be English or a local language used by the community. Researchers will explain to the volunteers on an individual basis, the nature of the study, what would be expected of them and their rights. Volunteers may choose to drop out of the study at any time without any restrictions. Volunteers will be informed that the screening procedure also includes physical examination and laboratory test. Following informed consent, using Consent to Participate Form (see attached) and counseling, volunteers may be enrolled for the study.

A baseline laboratory tests for: packed cell volume, white blood cell count with differentiation, platelet estimation, liver function (aspartate aminotransferase [SGOT], alanine aminotransferase [SGPT]), renal function (serum creatinine), blood urea nitrogen (BUN), pregnancy test (females only), HIV/AIDS, and hepatitis B and C tests will be done two weeks prior to dosing. Volunteers may not consume alcohol, tobacco, caffeine containing products, herbal or other drugs during the study.

Eligibility: The inclusion criteria are as follows: Adult males and females found normal on the basis of a pre-trial physical examination, medical history and the results of blood biochemistry and hematology tests; subject is competent and willing to sign informed consent form voluntarily after being given all the detailed information about the study; willingness to be hospitalized for a 24-hour intensive sampling period.

Exclusion criteria:

* Hypersensitivity to study drugs, alcoholism, anemia, evidence of pregnancy
* Abnormal laboratory test; smokers;
* Any clinically significant diseases or findings during the screening medical history or physical examination that, in the opinion of the investigator, may interfere with the study;
* Treatment with experimental or prescribed drugs within 30 days prior to the beginning of the study

Confidentiality: Volunteer's name as it appears on the questionnaire will be linked to an identification number. All other documents will have only the identification number instead of your name. The name will not be used in any public document. All written materials and consent forms will be stored in a locked file in the researcher's office. All materials will be destroyed by shredding five years after the completion of the research.

ELIGIBILITY:
Inclusion Criteria:

* The eligibility criteria included adults between 22 and 55 years;
* Healthy as determined on the basis of a pre-trial physical examination, medical history, electrocardiogram and the results of blood biochemistry and hematology tests;
* Subject was competent and willing to sign informed consent form voluntarily after being given all the detailed information about the study;
* Willing to be hospitalized for the 24-hour intensive sampling period.

Exclusion Criteria:

* The exclusion criteria was hypersensitivity to study drugs;
* Abnormal laboratory biochemistry values;
* Smokers;
* Any clinically significant diseases or findings during the screening, medical history or physical examination that, in the opinion of the investigator, may interfere with the study;
* Treatment with experimental drugs within 30 days prior to study entry.

Ages: 22 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2010-10; Primary Completion 2011-11 (Estimated); Study Completion 2011-12 (Estimated)

PRIMARY OUTCOMES:
Bioequivalence between the tests and reference drugs | 90 days
  The BE criterion established by the Food and Drug administration requires that the 90 % confidence interval of the ratio of suspension or tablet/co-administered liquid mixtures of the individual drugs for all the three parameters (Cmax, AUC0-t, AUC0-∞)should lie within 80 to 125 % range.

CONTACTS AND LOCATIONS:
Overall Officials: Moji C Adeyeye, Ph.D, Principal Investigator — Elim Pediatric Pharmaceuticals Inc. and Roosevelt University; Daniel A Gbadero, MD, Study Director — Bowen University Teaching Hospital, Ogbomoso, Nigeria
Locations (1):
- Bowen University Teaching Hospital, Ogbomoso, Oyo State, Nigeria

REFERENCES:
- [Background] Ellis JC, L'homme RF, Ewings FM, Mulenga V, Bell F, Chileshe R, Molyneux E, Abernethy J, van Oosterhout JJ, Chintu C, Walker AS, Gibb DM, Burger DM. Nevirapine concentrations in HIV-infected children treated with divided fixed-dose combination antiretroviral tablets in Malawi and Zambia. Antivir Ther. 2007;12(2):253-60. PMID 17503667